CLINICAL TRIAL: NCT04416854
Title: The Value of Palliative Primary Tumor Resection in Colon Cancer Patients With Initially Unresectable Metastases After Induction Chemotherapy: a Prospective, Multicenter, Randomized Controlled Clinical Trial
Brief Title: The Value of Palliative Primary Tumor Resection in Metastatic Colon Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, LI XIN-XIANG, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FDPRMCC
Record Dates: First submitted 2020-05-26; First posted 2020-06-04 (Actual); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Metastatic Colon Cancer; Surgery
Keywords: palliative surgery; stage IV colon cancer; chemotherapy
MeSH Terms: conditions — Colonic Neoplasms | interventions — XELOX

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Chemotherapy plus surgery (Experimental): Chemotherapy plus surgery: Four cycles of XELOX or six cycles of mFOLFOX6 combined with or without targeted therapy accroding to gene testing. After 4 cycles, the patients are randomized to surgery group. Patients receive palliative resection of Primary tumor. Then the rest four cycles XELOX or six cycles of mFOLFOX6 combined with or without targeted therapy are administrated.
  Interventions: Procedure: resection of primary tumor; Drug: XELOX; Drug: mFOLFOX6
- Chemotherapy alone (Active Comparator): Chemotherapy alone: Four cycles of XELOX or six cycles of mFOLFOX6 combined with or without targeted therapy accroding to gene testing. After 4 cycles, the patients are randomized to chemotherapy group. The rest four cycles XELOX or six cycles of mFOLFOX6 combined with or without targeted therapy are administrated.
  Interventions: Drug: XELOX; Drug: mFOLFOX6

INTERVENTIONS:
Procedure: resection of primary tumor — resection of primary lesion with unresectablely metastatic colon cancer
  Arms: Chemotherapy plus surgery
Drug: XELOX — Oxaliplatin 130mg/m2 ivgtt d1 and capecitabine 1000mg/m2,bid,po,d1-d14,every three weeks for a cycle
Drug: mFOLFOX6 — Oxaliplatin 85mg/m2, leucovorin 400mg/m2 ivgtt d1 and 5-FU 400 mg/m2 IV bolus d1，2400 mg/m2 CIV 46h, d1

SUMMARY:
The aim of this trial is to evaluate the value of palliative primary tumor resection in colon cancer patients with initially unresectable metastases and a positive response to induction chemotherapy which depends on gene testing. The primary endpoint is to evaluate overall survival.

ELIGIBILITY:
Inclusion Criteria:

* 75 years old
* ECOG (Eastern Cooperative Oncology Group) 0-1 and expected survival period for 6 months or more
* Pathological diagnosis of colon cancer adenocarcinoma
* At least one measurable objective tumor lesions which could be evaluated.
* Primary and metastatic tumors exist at the same time, and distant metastases are not resectable
* ANC≥1.5*109/L；PLT≥90*109/L；HB≥90g/L；TBI≤1.5(UNL); ALT、AST≤2.5ULN；Cr≤1.0(ULN) screening within 7 days
* No systemic chemotherapy
* Patients with voluntary participation, and sign the informed consent

Exclusion Criteria:

* Operation intervention required for perforation, bleeding and obstruction of intestinal cavity
* Multiple primary colorectal carcinoma
* Malignant peritoneal effusion or metastatic carcinoma of the peritoneum
* Uncontrolled pleural effusion
* Malignant tumour of the past five years with other organizations to source, but the full treatment of cervical carcinoma in situ and except skin basal cell carcinoma and squamous cell carcinomas
* With brain metastasis or meningeal metastasis
* Pregnancy or breast-feeding women
* Alcohol or drug addictions
* There is an important organ failure or other serious diseases, including coronary artery disease, symptomatic cardiovascular disease or myocardial infarction within 12 months; serious neurological or psychiatric history; severe infection; actively disseminated vascula blood coagulation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 627 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 5-year

SECONDARY OUTCOMES:
Progression-free survival 1 | 3-year
  The first progression time after diagnosis
Progression-free survival 2 | 3-year
  The first progression time after randomization
The rate of adverse events resulted from chemotherapy | 3-year
  The ratio of the number of patients experienced adverse events to the total patients
The quality of life postoperatively | 3-month, 6-month, 9-month, 12-month, 18-month, 24-month
  The European Organization for Research and Treatment (EORTC)-QLQ-C30 HRQL questionnaire was assessed with repeated measures at regular intervals postoperatively at months 3, 6, 9, 12, 18, and 24
Objective response rate | 1-year
The rate of postoperative complications | 1-year
  The ratio of the number of patients with postoperative complications to the total patients
The proportion of surgical intervention in control group | 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Center, Shanghai, Shanghai Municipality, China